CLINICAL TRIAL: NCT05419427
Title: A Randomized,Double Blind,Active Controlled Parallel Arm Multicenter Study Comparing Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Denosumab of Intas Pharmaceutical Limited (60 mg/mL) With Prolia® in Postmenopausal Women With Osteoporosis
Brief Title: Denosumab Biosimilar Injection in Post Menopausal Women With Osteoporosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lambda Therapeutic Research Ltd. (Industry)
Collaborators: Intas Pharmaceutical Limited (Biopharma Division) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0774-19; CTRI/2021/09/036190 (Registry Identifier: CTRI)
Record Dates: First submitted 2022-06-07; First posted 2022-06-15 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Denosumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: double-blinded. Participant, Investigator and Outcomes Assessor are masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Denosumab Solution for injection in single use prefilled syringe 60 mg permL (Experimental): Unit Dose Strength 60 mg per mL,Dosage Level 60 mg once every 6 months, Route of Administration-Subcutaneous injection
  Interventions: Drug: Denosumab
- Prolia® Solution for injection in single use prefilled syringe 60 mg per mL (Active Comparator): Unit Dose Strength 60 mg per mL,Dosage Level 60 mg once every 6 months,Route of Administration-Subcutaneous injection
  Interventions: Drug: Denosumab-Ref

INTERVENTIONS:
Drug: Denosumab — Denosumab 60 MG/ML
  Other Names: INTP23
  Arms: Denosumab Solution for injection in single use prefilled syringe 60 mg permL
Drug: Denosumab-Ref — Denosumab 60 MG/ML
  Other Names: Prolia
  Arms: Prolia® Solution for injection in single use prefilled syringe 60 mg per mL

SUMMARY:
Denosumab of Intas is biosimilar denosumab candidate under development by Intas Pharmaceutical Limited (Biopharma Division). Denosumab of Intas is already approved by Indian drug licensing authority- Drug Controller General (India) for marketing in Indian population since 2018.As per regulatory requirement, a comparative clinical study to establish Pharmacokinetic, Pharmacodynamic and Immunogenicity equivalence is required to conclude therapeutic equivalence to obtain marketing authorization of a biosimilar investigational product. This is a multicenter, randomized, double-blind, active controlled study in approximately 552postmenopausal women with osteoporosis.

An extension of the study is planned after completion of the initial 1 year of treatment. This extension is with the objective of submitting data on safety, and Immunogenicity, after switching of Prolia treatment arm to either Prolia or Intas denosumab for 6 months. This switching data is applicable only for FDA submission. Only patients who have undergone PK assessment will be eligible for the extension phase.

ELIGIBILITY:
Key Inclusion Criteria

* Participant must sign an ICF to participate in the study indicating that she understands the purpose of, and procedures required for the study as described in this protocol and is willing to and will be able to adhere to requirement of the protocol.
* Participant must be 55 to 90 years of age (both inclusive), at the time of signing the informed consent.
* Participants whose absolute bone mineral density T-score is less than equal to -2.5 and greater than equal -4.0 at the lumbar spine as measured by DXA (dual-energy x-ray absorptiometry), confirmed by the independent central imaging team
* At least two vertebrae in the L1-L4 region and at least one hip joint are evaluable by DXA, confirmed by the independent central imaging team.
* Postmenopausal ambulatory female and not considered to be of child-bearing potential if:

  a. Women are considered post-menopausal and not of child-bearing potential if, i. They have had 12 months of natural (spontaneous) amenorrhea (no vaginal bleeding or spotting) with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) OR ii. Six months of spontaneous amenorrhea with serum FSH levels greater than 40 mIU per mL OR iii. Have had surgical bilateral oophorectomy (with or without hysterectomy) at least six months ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment if she is considered not of child-bearing potential

Key Exclusion Criteria:

* Documented medical history of clinically significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Documented medical history of known allergies, hypersensitivity, or intolerance to denosumab or its excipients (refer to the IB)
* Documented medical history of metabolic or bone disease (except osteoporosis) that may interfere with the interpretation of the results, such as Pagets disease, osteomalacia, osteogenesis imperfecta, osteopetrosis, rheumatoid arthritis, ankylosing spondylitis or any other joint disease limiting mobility, Cushings disease, hyperprolactinemia, malabsorption syndrome
* Contraindications to the use of denosumab or Vitamin D and Calcium as per IB/local prescribing information at screening and/or baseline
* Documented medical history and/or current evidence of any of the following oral/dental conditions

  1. Prior history or current evidence of osteomyelitis or osteonecrosis of the jaw.
  2. Active dental or jaw condition which requires oral surgery.
  3. Planned invasive dental procedure expected during study period.
  4. Current evidence non-healed dental or oral surgery.
  5. Current evidence of poor oral hygiene
  6. Ill-fitting denture
* Current hyper- or hypocalcemia, defined as albumin-adjusted serum calcium outside the normal range at screening.
* Current, uncontrolled hyper- or hypoparathyroidism and history of hypoparathyroidism, per participant report or chart review. PTH outside the normal range (15-65 pg/mL) as assessed by central laboratory
* Current, uncontrolled hyper- or hypothyroidism, defined as thyroid stimulating hormone outside of the normal range (TSH-0.465 to 4.68 mIU/L) at screening.
* 25 (OH) Vitamin D lower than 20 ng/mL as assessed by the central laboratory at Screening. Vitamin D repletion will be permitted, and participants may be rescreened once.
* History and /or presence of 1 severe fracture or 2 moderate vertebral fractures
* Smokers or who have smoked within last 06 months prior to start of the study.
* Administration of bisphosphonate as follows: - c. IV Bisphosphonate in the past 3 years d. Oral bisphosphonates treatment for osteoporosis i. More than 3 years of cumulative use ii. Any dose received within 6 months prior to randomization iii. More than 1 month of cumulative use between 6 and 12 months prior to randomization
* Teriparatide or any PTH analogs treatment received within 12 months prior to randomization.
* Systemic oral or transdermal estrogen, SERMs, or calcitonin treatment of more than 1 month of cumulative use within 6 months prior to randomization.
* Androgen deprivation or hormonal ablation therapy of more than 1 month of cumulative use within 6 months prior to randomization.
* Tibolone or cinacalcet treatment received within 3 months prior to randomization
* Systemic glucocorticoids: Greater than equal to 5 mg prednisone equivalent per day for more than 10 days within 3 months prior to randomization.

Ages: 55 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 552 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2024-09-11 (Estimated); Study Completion 2024-11-24 (Estimated)

PRIMARY OUTCOMES:
Maximum measured concentration after first dose of denosumab and denosumab-ref., , | Day 1 to Day 181
Area under the concentration versus time curve from time zero to the last measurable concentration as calculated by linear trapezoidal method between denosumab and denosumab-ref postmenopausal women with osteoporosis | Day 1 to Day 181
Area under the concentration versus time curve from time zero to infinity. Where AUC 0-∞= AUC0-t + Ct2, Ct is the last measurable concentration and t2 is the terminal rate constant | Day 1 to Day 181

SECONDARY OUTCOMES:
Maximum percent reduction from baseline Emax percent reduction from baseline serum C-terminal telopeptide (CTX) after first dose of denosumab and denosumab-ref* | Day 1 to Day 181
Area under the percent reduction from baseline versus time curve from time zero to the last measurable concentration as calculated by linear trapezoidal method | Day 1 to Day 181

CONTACTS AND LOCATIONS:
Locations (1):
- S. R. Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/27/NCT05419427/Prot_000.pdf